CLINICAL TRIAL: NCT03440060
Title: Procalcitonin-guided Antibiotic Therapy During Severe Exacerbation of COPD Requiring Mechanical Ventilation: a Controlled Randomized Trial
Brief Title: Procalcitonin-guided Antibiotic Therapy During Severe Exacerbation of COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Mahdia (Other)
Responsible Party: Principal Investigator, Nejla Tilouche, principal investigator, University Hospital, Mahdia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301401
Record Dates: First submitted 2018-02-06; First posted 2018-02-20 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Acute Exacerbation Copd
Keywords: procalcitonin; mechanical ventilation; COPD exacerbation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard group (No Intervention): participants receive systematically empiric antibiotic therapy on admission with amoxicillin- acid clavulanic or levofloxacin in case of allergy
- Procalcitonin group (Active Comparator): participants receive antibiotics only if the procalcitonin value is at or greater than 0.25 ng/ml
  Interventions: Diagnostic Test: procalcitonin

INTERVENTIONS:
Diagnostic Test: procalcitonin — procalcitonin value will be obtained within 24 hours after ICU admission in both groups and will be taken into account in the procalcitonin group only
  Arms: Procalcitonin group

SUMMARY:
This study assess whether a procalcitonin guided antibiotic therapy can reduce significantly unnecessary antibiotic prescription during severe exacerbation of COPD requiring mechanical ventilation without compromising patients' outcome. The first group of patients will receive systematically empiric antibiotic therapy and the second group will receive antibiotics only if procalcitonin value is at or greater than 0.25 ng/ml.

DETAILED DESCRIPTION:
Recently, procalcitonin gained interest as the most reliable biomarker in predicting bacterial origin in low respiratory tract infections and sepsis.

Procalcitonin was shown to be non-inferior to standard guidelines in guiding antibiotic therapy during COPD exacerbation, without worsening patients' outcomes, and with a significant reduction in antibiotic exposure.

Its use to guide antibiotic treatment during COPD exacerbation may be more challenging because of the frequent colonization of the airways in patients with COPD, and thus it needs further evaluation.

Additionally, until today, no interventional studies evaluating procalcitonin protocol have been conducted in ventilated COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 40 years old who consent to the study protocol
* COPD diagnosis based on GOLD guidelines

Exclusion Criteria:

* Patients who did not consent
* Asthma
* Malignancy
* Immunocompromised
* Survival for at least 1 year is unlikely
* Patients already enrolled in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
time to recovery | 28 days
  defined by resolution of symptoms ( cough, sputum purulence and respiratory rate less than 25 breath per minute) and NIV withdrawal (normal pH for 24 consecutive hours after stopping NIV), for patients with home NIV investigators retain stabilization after returning to the same number of hours of NIV before current exacerbation and pH normalization for 24 consecutive hours

SECONDARY OUTCOMES:
Antibiotic exposure at day 90 | 90 days
  number of days the patient received antibiotics for any infection within 90 days from the day of admission
Hospital readmission for another exacerbation at day 90 | 90 days
  another readmission for another episode of COPD exacerbation within 90 days after a first discharge
NIV failure | 28 days
  clinical deterioration requiring invasive ventilation or death
ICU length of say (days) | 90 days
  number of days spent in the ICU during the index exacerbation
Hospital length of stay (days) | 90 days
  number of days spent in hospital during the index exacerbation
ICU mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tilouche Nejla, Mahdia, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathioudakis AG, Chatzimavridou-Grigoriadou V, Corlateanu A, Vestbo J. Procalcitonin to guide antibiotic administration in COPD exacerbations: a meta-analysis. Eur Respir Rev. 2017 Jan 31;26(143):160073. doi: 10.1183/16000617.0073-2016. Print 2017 Jan. PMID 28143877
- [Result] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Result] Schuetz P, Christ-Crain M, Thomann R, Falconnier C, Wolbers M, Widmer I, Neidert S, Fricker T, Blum C, Schild U, Regez K, Schoenenberger R, Henzen C, Bregenzer T, Hoess C, Krause M, Bucher HC, Zimmerli W, Mueller B; ProHOSP Study Group. Effect of procalcitonin-based guidelines vs standard guidelines on antibiotic use in lower respiratory tract infections: the ProHOSP randomized controlled trial. JAMA. 2009 Sep 9;302(10):1059-66. doi: 10.1001/jama.2009.1297. PMID 19738090